CLINICAL TRIAL: NCT01437384
Title: An Open-label, Single-sequence, Four-treatment Period Study to Evaluate Pharmacokinetic and Pharmacodynamic Interactions Between E5501 and Verapamil, and E5501 and Cyclosporine, Known P-glycoprotein Inhibitors in Healthy Subjects
Brief Title: Pharmacokinetic and Pharmacodynamic Study in Healthy Subjects Comparing the Interactions Between E5501 and Verapamil and Cyclosporine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E5501-A001-008
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Idiopathic Thrombocytopenic Purpura (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

ARMS (1):
- E5501 plus minus verapamil; plus minus cyclosporine (Experimental)
  Interventions: Drug: E5501

INTERVENTIONS:
Drug: E5501 — 20 mg oral dose of E5501; 240 mg once daily oral dose of sustained release verapamil; 400 mg oral dose of cyclosporine

SUMMARY:
36 healthy adult men and women will be enrolled with the goal of having 24 subjects complete the entire study. The study will consist of a pre-treatment phase and a treatment phase. The pre-treatment phase will include screening and baseline period 1. The treatment phase consists of 4 treatment period: Treatment Period 1 - administration of the first E5501 oral dose; Treatment Period 2 - administration of verapamil and the second E5501 oral dose; Treatment Period 3 - administration of the third E5501 dose; Treatment Period 4 - concomitant administration of cyclosporine and the fourth E5501 dose. A baseline period will precede each treatment period. The screening period will be up to 13 days in duration. After fulfilling screening requirements, subjects will check into the clinic on Day -1 for baseline assessments. They will be domiciled in the clinical testing facility for 6 days for Treatment Periods 1, 3, and 4 and will return intermittently for study procedures for 8 outpatient visits. They will be domiciled in the clinical testing facility for at least 14 days for Treatment Period 2 and will return intermittently for study procedures for 7 outpatient visits.

ELIGIBILITY:
Inclusion:

* Healthy adult men and women (age 18 to 55 years)
* Body mass index greater than or equal to 18kg/m2 and less than or equal to 32kg/m2 at the time of Screening and at each Baseline
* Platelet count between 120x109/L and 300x109/L at Baseline
* Women of childbearing potential must agree to use a highly effective method of contraception, other than estrogen-based hormonal contraceptives, during the treatment phase of the study

Exclusion:

* Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the PK of the study
* Agents associated with thrombotic events (including oral contraceptives) must be discontinued within 30 days of first study drug administration
* Evidence of organ dysfunction or any clinically significant event or illness in the subject's medical history, e.g., history of splenectomy
* History of arterial or venous thrombosis, including partial or complete thromboses (e.g., stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism). Known family history of hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency, etc.)
* Hemoglobin less than the lower limit of normal levels (women, 7.1 mmol/L; men, 8.1 mmol/L) In addition, other standard criteria for healthy volunteers will be used.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of E5501 | Periodically over the course of Days 1-11

SECONDARY OUTCOMES:
Platelet counts | Periodically over the course of Days 1-34

CONTACTS AND LOCATIONS:
Overall Officials: Gina Pastino, Study Director — Eisai Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States